CLINICAL TRIAL: NCT02326727
Title: Influence of Epidural Analgesia on Natural Killer Cell (NK) Activity After Colonic Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0095-14-HYMC
Record Dates: First submitted 2014-12-10; First posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Colonic Neoplasms
Keywords: Epidural Analgesia; Natural Killer Cells
MeSH Terms: conditions — Colonic Neoplasms | interventions — Ropivacaine; Fentanyl; Propofol; Isoflurane; Nitrous Oxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Anesthesia (Active Comparator): Patients receiving general anesthesia with Fentanyl,Propofol, Isoflurane and Nitrous Oxide only during colonic cancer surgery
  Interventions: Drug: Fentanyl; Drug: Propofol; Drug: Isoflurane; Drug: Nitrous Oxide
- Combined anesthesia (Active Comparator): Patients receiving general anesthesia and epidural analgesia with Ropivacaine during colonic cancer surgery
  Interventions: Drug: Ropivacaine; Drug: Fentanyl; Drug: Propofol; Drug: Isoflurane; Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Ropivacaine — Epidural analgesia
  Arms: Combined anesthesia
Drug: Fentanyl — General Anesthesia
Drug: Propofol — General Anesthesia
Drug: Isoflurane — General Anesthesia
Drug: Nitrous Oxide — General Anesthesia

SUMMARY:
Regional anesthesia may decrease the release of endogenous opioids, increase Natural Killer cell (NK) function and decrease development of metastasis. The recent analysis of the Cancer Registry has noted an improved 5-year survival in patients who received epidural analgesia during surgery for colorectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonic cancer surgery

Exclusion Criteria:

* Patients with poor physical status Patients needed emergency surgery Coagulopathic disorders with international normalized ratio (INR) level more than 1.4 Thrombocytopenia with platelets count less 100000 per mcl Allergic reaction to local anesthetics in patient history Failure to performing the epidural analgesia from another cause Preoperative immunomodulating treatment Recent history of chemotherapy or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Count of live and dead target erythroleukemic cells | 72 hours
  All clinical and laboratory parameters from blood samples taken before and after the operation will be compared between the two groups of patients. The nominal data comparison will be performed by ANOVA test, and the nonparametric data will be performed by Mann-Whitney test and interquartile ranges (IQR) for non-normally distributed data.
Plasma concentration of cytokines | 72 hours
  All clinical and laboratory parameters from blood samples taken before and after the operation will be compared between the two groups of patients. The nominal data comparison will be performed by ANOVA test, and the nonparametric data will be performed by Mann-Whitney test and interquartile ranges (IQR) for non-normally distributed data.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel